CLINICAL TRIAL: NCT07008820
Title: Patient Reported Outcomes and Patient Voice Among Patients Diagnosed With Low Risk Myelodysplastic Syndrome (LR-MDS) or Unexplained Anemia In Japan
Status: Recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA056-1133
Record Dates: First submitted 2025-05-27; First posted 2025-06-06 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Myelodysplastic Syndrome (MDS)
Keywords: Myelodysplastic Syndrome (MDS)
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Low Risk Myelodysplastic Syndrome erythropoietin stimulating agent naïve and non-transfusion dependent
  Interventions: Other: Health-related quality of life questionnaires; Other: Qualitative interviews
- Cohort 2: Suspected Low Risk Myelodysplastic Syndrome with unexplained anemia
  Interventions: Other: Health-related quality of life questionnaires; Other: Qualitative interviews

INTERVENTIONS:
Other: Health-related quality of life questionnaires — Questionnaires include:
  EORTC-QLQ C30 FACT-An PGI-S EQ-5D-5L
Other: Qualitative interviews — For participants that meet eligibility criteria

SUMMARY:
This study will examine quality of life, experiences, and unmet needs among individuals diagnosed with Low Risk Myelodysplastic Syndrome who are erythropoietin stimulating agent naïve and non-transfusion dependent and among individuals with suspected myelodysplastic syndromes with unexplained anemia in Japan

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria for the quantitative phase will include either 1 or 2 and all of 3-6:

1. Low Risk Myelodysplastic Syndromes (LR MDS) erythropoietin stimulating agent (ESA) naïve non-transfusion dependent (NTD) patrticipants: identified with confirmed via bone marrow aspirate and < 5% blasts in bone marrow. Lower-risk is defined by International Prognostic Scoring System (IPSS) or Revised International Prognostic Scoring System (IPSS-R), as follows:

   * Very low, low, or intermediate-risk (score ≤ 3.5) as assessed by IPSS-R
   * Low or intermediate-1 (score ≤ 1) as assessed by IPSS
2. Unexplained anemia with suspected MDS: identified anemia with general anemia (iron/vitamin deficiency, bleeding, renal, etc.) excluded
3. Participants with hemoglobin in the most recent blood test < 10.0 g/dl, or the average of hemoglobin < 10.0g/dl in the most recent 2 blood tests conducted within 30 days prior to enrollment in this study
4. Participants who are ≥ 18 years of age at the time of signing the informed consent form.
5. Participants who are able and willing to provide informed consent.
6. Participants who are able to complete the protocol requirements.

For the qualitative phase (approximately 10 participants), the inclusion criteria will also include:

1. Participants with severity scores of "moderate" or greater on at least one Patient Global Impression-Severity (PGI-S) item.

Exclusion Criteria:

Patients meeting the following criteria will be excluded:

1. Participants who have difficulty obtaining informed consent or execution of this study because of insufficient Japanese language proficiency.
2. Participants who are considered to have difficulty answering HRQoL questionnaires and/or responding to questions during cognitive interview
3. Participants who received red-blood cell transfusion (RBC-T) within 16 weeks prior to enrollment.

   Note: RBC-T of 1 to 2 units within the 16 weeks prior to enrollment are allowed, provided those 1-2 RBC-T units are administered for an acute event/illness (i.e., surgical procedure, bleeding, infection) or presence of comorbidity (including cardiovascular, pulmonary, cerebrovascular), and not for the treatment of low hemoglobin (with or without symptoms) alone.
4. Participants who received prior drug treatment related to anemia; drugs include the following: erythropoiesis stimulating agent, erythroid maturation agent, hypomethylating agent, immunomodulatory drugs, immuno-suppressive agent.
5. Participants with myelodysplastic/myeloproliferative neoplasms (MDS/MPN) according to World Health Organization (WHO) 2016 classification (i.e., chronic myelomonocytic leukemia, atypical chronic myeloid leukemia, breakpoint cluster region-Abelson 12, juvenile myelomonocytic leukemia, MDS/MPN unclassifiable).
6. Participants with secondary MDS (i.e., MDS that is known to have arisen as a result of chemical injury or treatment with chemotherapy and/or radiation for other diseases).
7. Participants with a known history of diagnosis of acute myeloid leukemia.
8. Participants with major surgery within 8 weeks prior to enrollment. Patients must have completely recovered from any previous surgery prior to enrollment.
9. Participants with history of cerebrovascular accident (including ischemic, embolic, and hemorrhagic cerebrovascular accident), transient ischemic attack, deep venous thrombosis (including proximal and distal), pulmonary or arterial embolism, arterial thrombosis, or other venus thrombosis within 6 months prior to enrollment. Note: prior superficial thrombophlebitis is not an exclusion criterion.
10. Participants who have any condition or receive concomitant medication that confounds the ability to interpret data from the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include adult participants diagnosed with Low Risk Myelodysplastic Syndrome who are erythropoietin stimulating agent naïve and non-transfusion dependent or adults with suspected myelodysplastic syndromes with unexplained anemia in Japan
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Participant quality of life as assessed by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC-QLQ C30) patient reported outcome questionnaire | Day 1
Participant anemia symptoms as assessed by the Functional Assessment of Cancer Therapy - Anemia (FACT-An) patient reported outcome questionnaire | Day 1
Symptom severity as assessed by the Patient Global Impression-Severity (PGI-S) patient reported outcome questionnaire | Day 1
General health status of participants as assessed by the EQ-5D-5L patient reported outcome questionnaire | Day 1
Participant baseline socio-demographics | Baseline
Participant baseline clinical characteristics | Baseline

SECONDARY OUTCOMES:
Qualitative interview results | Up to 1 month
  Qualitative interview questions to include questions to understand the participants:
  * Experiences of diagnosis and treatment
  * Symptoms of anemia
  * Quality of life
  * Communication with physicians
  * Satisfaction with current treatments

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Mebix. Inc, Minato-ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts